CLINICAL TRIAL: NCT01360619
Title: Clinical Study About Fat Measurement on Multifunction Keito by Comparison Versus Its Predicate K014009
Status: Completed | Type: Observational
Sponsor: Aguiflai Iberica, S.L. (Industry)
Responsible Party: Angel Pons ferre, Aguiflai Iberica, S.L.
Other Study IDs: K8-FAT-05062007
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2007-10

CONDITIONS: Body Fat
Keywords: To demonstrate that multifunction Keito is as effective, as safe and accurate as the predicate K014009 on its body fat measurement.

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The researchers believe that the multifunction Keito devices shares with TANITA TBF-300 (K014009) the same efficacy on the body fat measurement. Even if the body contact points are not the same, the researchers deeply believe that the tetrapolar BIA used by the predicate gives results as similar as the multifunction keito does.

DETAILED DESCRIPTION:
177 volunteers were enrolled in this clinical Study. Before taking the fat measurement by the devices under test, the observers measured the weight and height of each volunteer prior to measure the body fat. This was done to configure a preliminary idea about the body composition of the subject.

Both devices are designed by the same technology to emit a low current through the body, and finally make a measurement of the impedance found between the body contact points. We expected the results to be very similar.

ELIGIBILITY:
Inclusion Criteria:

* All population who meet with the requirements described on the user's manual.

Exclusion Criteria:

* Pregnant women.
* Individuals who have a pacemaker or any other internal medical device.
* Population whose weight is under 15 Kg and less than 135 cm tall.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To include the maximum types of patients, the selection was opened to all the general public who could use the multifunction Keito in a public site, where is is intended to be placed. The test was carried out following the user's manual rules about who can use the device.
Sampling Method: Probability Sample
Enrollment: 177
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Angel P Ferre, Telecommunications Engineer, Principal Investigator — Aguiflai Iberica, S.L.
Locations (1):
- Aguiflai Iberica, s.l, Vilassar de Mar, Barcelona, Spain